CLINICAL TRIAL: NCT05331625
Title: Understanding Quality of Life Among Patients With Cancer Receiving Palliative Care
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Scott Halpern, Associate Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UPCC 11922; 850807 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2022-04-01; First posted 2022-04-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-02

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants in this group will consent to participate in a study about quality of life for patients with cancer seeking outpatient palliative care. They will be seen in a palliative care oncology clinic at which time they will be offered additional resources to promote symptom management. They will be asked to complete a series of surveys every two weeks for 16 weeks which will assess their quality of life, symptoms, and medication use.
  Interventions: Behavioral: Offering Additional Resources to Promote Symptom Management
- Usual Care (No Intervention): Participants in this group will consent to participate in a study about quality of life for patients with cancer seeking outpatient palliative care. They will be seen in a palliative care oncology clinic where they will receive symptom management and supportive care. They will be asked to complete a series of surveys every two weeks for 16 weeks which will assess their quality of life, symptoms, and medication use.

INTERVENTIONS:
Behavioral: Offering Additional Resources to Promote Symptom Management — Participants will be offered additional resources to promote symptom management.
  Arms: Intervention

SUMMARY:
This randomized controlled trial will assess the effects on quality of life of two approaches to symptom management among new patients referred to a palliative care oncology clinic.

ELIGIBILITY:
Inclusion Criteria:

* Be a new patient at an outpatient palliative care clinic
* Resident of Pennsylvania
* Over 18 years of age

Exclusion Criteria:

* Prior use of certain symptom focused therapies
* Currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Quality of Life - McGill Quality of Life Questionnaire | Baseline - 16 weeks
  Quality of life will be measured through the McGill Quality of Life Questionnaire Revised (MQOL-R). The questionnaire is 15 questions assessing overall and specific areas of quality of life.

SECONDARY OUTCOMES:
Feasibility of Accessing Additional Resources for Symptom Management | Baseline - 16 weeks
  Feasibility will be measured by whether participants accessed the additional resources for symptom management.
Acceptability of Accessing Additional Resources for Symptom Management | Baseline - 16 weeks
  Acceptability will be measured by whether participants accessed the additional resources for symptom management.
Symptom Severity | Baseline - 16 weeks
  Symptom severity will be measured through the Edmonton Symptom Assessment System (ESAS). The survey is 10 questions assessing the severity of pain, nausea, depression, etc. on a 0 to 10 scale-in which a 0 representing best possible state/symptom absence and a 10 representing worst possible state.
Medication Use | Baseline - 16 weeks
  Medication use will be measured through a medication diary created for the study. The medication diary asks participants about recent medications, amounts, and dosages.
Hospital-Free Days | Baseline - 16 weeks
  Hospital-free days will be measured through examination of participant's electronic health record.
Mortality | Baseline - 16 weeks
  Mortality will be measured through examination of participant's electronic health record.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No